CLINICAL TRIAL: NCT00698451
Title: A Phase II Single Arm Study of Carboplatin and DOXIL (PLD) Plus Bevacizumab in Patients With Platinum Sensitive Recurrent Ovarian, Fallopian Tube and Primary Peritoneal Cancers
Brief Title: A Study of Carboplatin and DOXIL Plus Bevacizumab in Patients With Platinum Sensitive Recurrent Ovarian, Fallopian Tube and Primary Peritoneal Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Centocor Ortho Biotech Services, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015094; DOXILOVC2007 (Other: Johnson & Johnson Pharmaceutical Research and Development)
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Results first posted 2013-07-12 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-08

CONDITIONS: Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms
Keywords: Ovarian cancer; fallopian tube cancer; primary peritoneal cancer; DOXIL; carboplatin; bevacizumab
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — Bevacizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): doxorubicin HCL liposome; bevacizumab; carboplatin30 mg/m2 by intravenous infusion Day 1 of each 28 day cycle; 10 mg/kg by intravenous infusion Days 1 and 15 of each 28 day cycle; AUC=5 by intravenous infusion Day 1 of each 28 day cycle
  Interventions: Drug: doxorubicin HCL liposome; bevacizumab; carboplatin

INTERVENTIONS:
Drug: doxorubicin HCL liposome; bevacizumab; carboplatin — 30 mg/m2 by intravenous infusion Day 1 of each 28 day cycle; 10 mg/kg by intravenous infusion Days 1 and 15 of each 28 day cycle; AUC=5 by intravenous infusion Day 1 of each 28 day cycle

SUMMARY:
The purpose of this study is to evaluate the response rate (Complete Response (CR) and Partial Response (PR)) to carboplatin and DOXIL treatment in combination with bevacizumab in patients with platinum-sensitive recurrent ovarian, fallopian tube and primary peritoneal cancers. All patients will received DOXIL, carboplatin and bevacizumab for a maximum of ten 28-day cycles. Patients will be followed for six months following treatment to assess progression-free survival.

DETAILED DESCRIPTION:
DOXIL pegylated liposomal doxorubicin (PLD) is approved for use in patients with ovarian cancer whose disease has progressed or recurred after platinum-based chemotherapy. Data suggest that combination therapy of carboplatin plus DOXIL provides superior benefit to single agent therapy. Bevacizumab, a vascular endothelial growth factor (VEGF) inhibitor, is approved for use in combination with intravenous 5-fluorouracil-based chemotherapy for the treatment of metastatic colorectal cancer and in combination with carboplatin and paclitaxel (treatment of non-small cell lung cancer); and with paclitaxel (first line treatment of metastatic HER2-negative breast cancer). There are data showing bevacizumab has activity in the treatment of ovarian cancer, and it is currently being studied in platinum-sensitive relapsed ovarian cancer in combination with carboplatin/gemcitabine. No data exist on the efficacy and safety of bevacizumab administered with carboplatin and DOXIL. Based on the growing interest of incorporating bevacizumab in to ovarian cancer treatment and the activity seen to date, the evaluation of the combination of carboplatin and DOXIL with bevacizumab is warranted. This is a single arm (one dosing regimen), multicenter, open label (both the patient and the physician know what drug is being given) study in patients with platinum-sensitive recurrent ovarian, fallopian tube or primary peritoneal cancers. This study will be conducted in multiple sites across the United States. All patients will receive DOXIL, carboplatin and bevacizumab by intravenous (IV) infusion for a maximum of ten (10) 28-day cycles. A disease response assessment will occur after the completion of Cycles 2, 4, 6, 8 and at the end of treatment. Patients will be followed for six (6) months post-treatment for progression-free survival. Disease progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST). RECIST is an accepted classification for response to treatment with classifications of Complete Response (CR), Partial Response( (PR), Progressive Disease (PD) or Stable Disease (SD).The primary objective of this study is to evaluate the objective response rate (Complete Response (CR) and Partial Response (PR)) to carboplatin and DOXIL treatment in combination with bevacizumab in patients with platinum-sensitive recurrent ovarian, fallopian tube and primary peritoneal cancers. The secondary objectives are to assess the safety profile of carboplatin and DOXIL in combination with bevacizumab as well as the following efficacy endpoints: Duration of response, Progression-free Survival, and Time to Progression. Safety will be evaluated using adverse events, clinical laboratory tests, and tests for cardiac function after the first 20 patients have been entered and received at least 2 cycles of therapy. Overall safety will be summarized at study completion. DOXIL (30 mg/m2), and carboplatin (area under the curve (AUC 5)) will be given on Day 1 of each 28-day cycle. Bevacizumab (10 mg/kg) will be given on days 1 and 15 of every 28-day cycle. All treatment will be given by intravenous (IV) infusion and repeated every 4 weeks for up to 10 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of epithelial ovarian, fallopian tube or primary peritoneal cancer
* Relapse-free interval of >6 months afer completion of first line platinum-based chemotherapy
* Measurable disease (at least one lesion that can be accurately measured in a least 1 dimension)
* Adequate bone marrow function, renal, and liver function. Normal cardiac function
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

Exclusion Criteria:

* No patients who have received more than 1 previous regimen of chemotherapy (maintenance is not considered a second regimen)
* No patients receiving immunotherapy or radiotherapy or patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis
* No patients who require parenteral hydration or nutrition or have clinical signs or symptoms of gastrointestinal bowel obstruction or perforation
* No patients with previous or current malignancy other than basal cell or squamous cell carcinoma of the skin
* No patients with clinically significant cardiovascular disease
* No patients with a history of bevacizumab or other VEGF or VEGF receptor-targeted agent use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McGowan, MD, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Horsham, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DOXIL/CARBOPLATIN/BEVACIZUMAB: Doxorubicin HCL liposome; bevacizumab; carboplatin30 mg/m2 by intravenous infusion Day 1 of each 28 day cycle; 10 mg/kg by intravenous infusion Days 1 and 15 of each 28 day cycle; AUC=5 by intravenous infusion Day 1 of each 28 day cycle Intervention.
Period: Overall Study
Arm/Group | DOXIL/CARBOPLATIN/BEVACIZUMAB
Started | 54
Completed | 15
Not Completed | 39
Not completed — Adverse Event | 22
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 6
Not completed — Withdrawal by Subject | 6
Not completed — Disease progression | 3

BASELINE CHARACTERISTICS:
Arm/Group | DOXIL/CARBOPLATIN/BEVACIZUMAB
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy End Point is the Number of Patients With an Objective Response.
Description: Objective Response Rate to Treatment is defined as the Proportion of Patients With a Complete Response (CR) or Partial Response (PR). A Complete Response (CR) is the disappearance of all target lesions and a Partial Response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD
Time Frame: Approximately 280 days (from start of treatment to the end of 10 cycles of treatment where each cycle is 28 days)
Population: ITT
Measure: Number; unit: Participants
Groups:
- DOXIL/CARBOPLATIN/BEVACIZUMAB: doxorubicin HCL liposome; bevacizumab; carboplatin30 mg/m2 by intravenous infusion Day 1 of each 28 day cycle; 10 mg/kg by intravenous infusion Days 1 and 15 of each 28 day cycle; AUC=5 by intravenous infusion Day 1 of each 28 day cycle
Arm/Group | DOXIL/CARBOPLATIN/BEVACIZUMAB
Number analyzed (Participants) | 54
Participants | 39
Statistical Analysis 1: Comparison: DOXIL/CARBOPLATIN/BEVACIZUMAB; Test type: Superiority or Other; p = 0.05, Exact Binomial Distribution; Percentage = 72.2, 95% CI 2-sided [58.4 to 83.5]

2. Secondary Outcome: The Secondary Efficacy Endpoints is Duration of Objective Response.
Description: Objective Response Rate to Treatment Defined as the Proportion of Patients With a Complete Response (CR) or Partial Response (PR) Where a Complete response (CR) is the disappearance of all target lesions and a Partial Response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Duration of response: Duration of response was defined only for subjects with CR or PR as the best overall response. It was calculated from the date of first documentation of response to the date of disease progression or death due to progressive disease.
Time Frame: Duration of response was defined only for subjects with CR or PR as the best overall response. It was calculated from the date of first documentation of response to the date of disease progression or death due to progressive disease.
Population: ITT
Measure: Median (Full Range); unit: Days
Arm/Group | DOXIL/CARBOPLATIN/BEVACIZUMAB
Number analyzed (Participants) | 54
Days | 362 [282 to NA] — Duration of response was defined only for subjects with CR or PR as the best overall response. It was calculated from the date of first documentation of response to the date of disease progression or death due to progressive disease.

ADVERSE EVENTS:
Arm/Group | DOXIL/CARBOPLATIN/BEVACIZUMAB
Serious Adverse Events (participants affected / at risk) | 15/54
Other Adverse Events (participants affected / at risk) | 53/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOXIL/CARBOPLATIN/BEVACIZUMAB (N=54)
Constipation (Gastrointestinal disorders) | 1 (1)
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Small Intestinal Perforation (Gastrointestinal disorders) | 1 (1)
Abdominal Abscess (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 1 (1)
Corneal Abrasion (Injury, poisoning and procedural complications) | 1 (1)
Device Malfunction (Injury, poisoning and procedural complications) | 1 (1)
Device Occlusion (Injury, poisoning and procedural complications) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Ureteric Obstruction (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOXIL/CARBOPLATIN/BEVACIZUMAB (N=54)
Fatigue (General disorders) | 32 (32)
Mucosal Inflammation (General disorders) | 8 (8)
Chest Pain (General disorders) | 7 (7)
Oedema Peripheral (General disorders) | 6 (6)
Pain (General disorders) | 5 (5)
Pyrexia (General disorders) | 5 (5)
Feeling Hot (General disorders) | 3 (3)
Oedema (General disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 31 (31)
Stomatitis (Gastrointestinal disorders) | 20 (20)
Diarrhoea (Gastrointestinal disorders) | 18 (18)
Vomiting (Gastrointestinal disorders) | 16 (16)
Constipation (Gastrointestinal disorders) | 15 (15)
Abdominal Pain (Gastrointestinal disorders) | 12 (12)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (4)
Flatulence (Gastrointestinal disorders) | 4 (4)
Dry Mouth (Gastrointestinal disorders) | 3 (3)
Gingival Bleeding (Gastrointestinal disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 28 (28)
Thrombocytopenia (Blood and lymphatic system disorders) | 28 (28)
Neutropenia (Blood and lymphatic system disorders) | 23 (23)
Leukopenia (Blood and lymphatic system disorders) | 20 (20)
Headache (Nervous system disorders) | 23 (23)
Dizziness (Nervous system disorders) | 13 (13)
Peripheral Sensory Neuropathy (Nervous system disorders) | 6 (6)
Dysgeusia (Nervous system disorders) | 5 (5)
Neuropathy Peripheral (Nervous system disorders) | 4 (4)
Memory Impairment (Nervous system disorders) | 3 (3)
Sinus Headache (Nervous system disorders) | 3 (3)
Syncope (Nervous system disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 28 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 15 (15)
Rash (Skin and subcutaneous tissue disorders) | 13 (13)
Dry Skin (Skin and subcutaneous tissue disorders) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 11 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (7)
Decreased Appetite (Metabolism and nutrition disorders) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 6 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Hypertension (Vascular disorders) | 20 (20)
Flushing (Vascular disorders) | 6 (6)
Hot Flush (Vascular disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 20 (20)
Haematuria (Renal and urinary disorders) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 8 (8)
Anxiety (Psychiatric disorders) | 6 (6)
Depression (Psychiatric disorders) | 6 (6)
Urinary Tract Infection (Infections and infestations) | 8 (8)
Nasopharyngitis (Infections and infestations) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3)
Neutrophil Count Decreased (Investigations) | 5 (5)
Weight Decreased (Investigations) | 4 (4)
Palpitations (Cardiac disorders) | 4 (4)
Tachycardia (Cardiac disorders) | 4 (4)
Vision Blurred (Eye disorders) | 5 (5)
Hypersensitivity (Immune system disorders) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days